CLINICAL TRIAL: NCT04606186
Title: Influence of Probiotics on Clinical Parameters, the Oral Microbiome and the Immune System During an Orthodontic Treatment in Adult Patients: a Prospective, Double-blind, Randomized, Clinical Study
Brief Title: Influence of Probiotics on Clinical Parameters, the Oral Microbiome and the Immune System During an Orthodontic Treatment in Adult Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Erlangen-Nürnberg (Other)
Collaborators: BioGaia AB (Industry)
Responsible Party: Principal Investigator, Dr. Corinna Lesley Seidel, Orthodontist, University of Erlangen-Nürnberg
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ER-Ortho-Pro-RCT-Erw-2
Record Dates: First submitted 2020-09-09; First posted 2020-10-28 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Gingivitis; Periodontal Inflammation; Orthodontic Appliance Complication
Keywords: Orthodontics; Inflammation; Microbiome; Probiotics
MeSH Terms: conditions — Gingivitis; Inflammation

STUDY DESIGN:
Intervention Model Description: Monocentric, randomized, double-blind, placebo-controlled, clinical study
Who Masked: Participant, Investigator
Masking Description: Study participants, meeting the inclusion criteria and not fulfilling the exclusion criteria, will be assigned to the study group or to the control group using a randomization plan. Randomization plan will be generated by the Center for Clincal Studies of the University Hospital of Erlangen. The lab manager will prepare storage boxes, in which exactly 168 lozenges will be stored. Half of the boxes will contain test-lozenges (study group), half or them will contain placebo-lozenges (control group). The storage boxes for the test and the placebo group will be identical and blinded. The storage boxes will be labelled with pseudonyms in accordance to the randomization plan generated by the Center for Clinical Studies. Therefore, study participants will not have knowledge of the group affiliation. The collection of the samples and the measuring of the clinical parameters will be performed by one orthodontist, who will be blinded to the randomization of the study participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lactobacillus reuteri Prodentis®-lozenges (Active Comparator)
  Interventions: Dietary Supplement: Lactobacillus reuteri Prodentis®-lozenges (DSM 17938, ATCC PTA 5289)
- Placebo-lozenges (BioGaia) (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo-lozenges (BioGaia)

INTERVENTIONS:
Dietary Supplement: Lactobacillus reuteri Prodentis®-lozenges (DSM 17938, ATCC PTA 5289) — Supplementary intake of Lactobacillus reuteri Prodentis®-lozenges (DSM 17938, ATCC PTA 5289) 2 times per day for 12 weeks
  Arms: Lactobacillus reuteri Prodentis®-lozenges
Dietary Supplement: Placebo-lozenges (BioGaia) — Placebo-lozenges (BioGaia)
  Arms: Placebo-lozenges (BioGaia)

SUMMARY:
Orthodontic treatment with fixed appliances can be necessary to correct malocclusions in adolescence or adulthood. It its known that orthodontic treatment induces aseptic pseudo-inflammatory reactions. However, studies could show that an increase of certain inflammatory cytokines during orthodontic treatment correlated with a higher risk of root resorption. Moreover, it has been shown that orthodontic treatment leads to a dysbiosis of the oral microbiome especially during the first 3 months of the orthodontic treatment. This could be a potential risk factor as the inflammation of periodontitis during an orthodontic treatment could favor root resorption and progressive destruction of the periodontal apparatus.

Probiotics are already used successfully as an adjuvant therapy in the treatment of periodontitis to improve clinical parameters and to reduce local inflammation. However, there are only a few studies that investigated the influence of probiotics during an orthodontic treatment.

Therefore, the aim of our study is to investigate if the daily intake of lozenges containing probiotics versus placebo lozenges during the first 3 months of orthodontic treatment with fixed appliances can improve clinical parameters, reduce local inflammation, systemic inflammation and prevent a dysbiosis of the oral microbiome.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years and older) with fixed appliances undergoing orthodontic treatment.
* Signed declaration of consent by the patient

Exclusion Criteria:

* • Systemic or metabolic disease that are related to gingivitis or (e.g. diabetes) or could possibly influence the oral microbiome

  • obesity:
* body mass index (BMI) > 30 kg/m² (weight and height will be measured)

  • Eating disorder or underweight
* BMI < 18,5 kg/m² (weight and height will be measured)

  * Above-average consumption of milk products: > 3 portions/day = >1,2 liters of milk or 1200g yoghurt/day (daily dose recommended by the german society for nutrition = 1-3 portions of milk products)
  * allergy to ingredients of the lozenges
  * intake of antibiotics or dietary supplementation (probiotics, vitamin C/D) in the last 6 months or during the study
  * regular use of antibacterial mouth wash
  * pregnancy
  * smoking
  * retraction of the declaration of consent by the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2020-10-19 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Gingival Index (GI) | Baseline to week 4 of intake
  Primary endpoint is the change of the Gingival Index (GI) from baseline to week 4. The measurement of GI is described by Löe et al, which scores the gingival condition according to the defined criteria. The scores will be measured at four sites per tooth, added and divided by four to obtain the "GI for the tooth"-Index. We will use the 'GI for the tooth' described there, but only for those teeth with fixed ortodontic brackets. The 'GI for the patient' is then the mean of the GIs for the teeth.
  CRITERIA FOR THE GINGIVAL INDEX SYSTEM
  0 = Absence of inflammation.
  1. = Mild inflammation - slight cliange in color and little change in texture.
  2. = Moderate inflammation - modcrate glazing, redness,oedema, hypertrophy, bleeding on pressure.
  3. = Severe inflammation - marked redness and hypertrophy, tendency to spontaneous bleeding, ulceration.

SECONDARY OUTCOMES:
Probing pocket depth (PPD) (4-point-measurement) | Baseline till 12 months after insertion of appliance
  The measurement of the probing of periodontal pockets (periodontal probing depth, PPD) is performed according to standardized protocols: insertion of a perdiotonal probe into the gingival sulcus with a force of 0.2-0.3 N; probing depth is read out at landmarks on the periodontal prove. The scores will be measured at four sites per tooth, added and divided by four to obtain the "PPDI for the tooth"-Index. We will use the 'PPD for the tooth', but only for those teeth with fixed ortodontic brackets. The 'PPD for the patient' is then the mean of the PPDs for the teeth.
Modified Plaque Index (MPI) | Baseline till 12 months after insertion of appliance
  The measurement of Modified plaque index (MPI) is described by Attin et al, which scores the amount of plaque according to the defined criteria. The score will be measured at each tooth, but only for those teeth with fixed ortodontic brackets. The 'Modified plaque index for the patient' is then the mean of the MPIs per teeth: Index = (Sum of MPI per tooth×100)/ (3×number of measured teeth).
  CRITERIA FOR THE MODIFIED PLAQUE INDEX
  0 = no plaque
  1. = small plaque areas approximal
  2. = small plaque areas approximal + cervical
  3. = plaque covers 1/3 of the cervical area of the bracket.
Local cytokine expression | Baseline till 12 months after insertion of appliance
  Samples from different oral niches (saliva, soft and hard tissue samples, gingival crevicular fluid) will be collected to analyse local inflammation: Unstimulated saliva will be gained by the spitting method, soft tissue samples will be collected in using sterile swabs, hard tissue samples of supragingival plaque will taken by sterile curettes and samples of gingival sulcus fluid will be collected from 6 periodontal pockets of the mesio-buccal side of defined teeth (Ramfjord teeth: 16,21,24,36,41,44) using sterile paper strips. Sulcus fluid flow rate will be performed using Periotron 8000. The cytokine concentration (in pg/mL) of granulocyte-macrophage colony-stimulating-factor (GM-CSF), interferon (IFN)- gamma, interleukin (IL)-2, IL-4, IL-6, IL-8 and IL-10 as well as tumor necrosis factor (TNF) in defined oral niches will be measured using multiplex immunoassay.
Oral microbiome | Baseline till 12 months after insertion of appliance
  Samples from different oral niches (saliva, soft and hard tissue samples, gingival crevicular fluid) will be collected to analyse the oral microbiome: Unstimulated saliva will be gained by the spitting method, soft tissue samples will be collected in using sterile swabs, hard tissue samples of supragingival plaque will taken by sterile curettes and samples of gingival sulcus fluid will be collected from 6 periodontal pockets of the mesio-buccal side of defined teeth (Ramfjord teeth: 16,21,24,36,41,44) using sterile paper strips. Composition of the oral microbiome will be analysed using 16 S rRNA sequencing and operational taxonomic units (OTUs) will be classified according to SILVA database.
Systemic cytokine expression | Baseline till 12 months after insertion of appliance
  Samples of peripheral whole blood will be taken. Measurement of systemic cytokine concentration in serum (in pg/mL) will be performed using Enzyme-linked immunosorbent assay (ELISA). To analyse systemic inflammation and a possible Th1-/Th2- or Th-17 shift, cytokines representing the Th1-/Th-2/Th-17 cytokine profile (e.g. TNF, Interferon-Gamma,Interleukin 10) will be measured.
Cellular immunity | Baseline till 12 months after insertion of appliance
  Samples of peripheral whole blood will be taken.Composition of immunoregulatory cells in the mononuclear cell fraction (MNC) will be analysed using samples of peripheral blood and MNC isolation. The cellular immune status will be analysed quantitatively (in %: relative percentual distribution in the MNC fraction) using fluor-activated cell scanning (FACS). Lymphocyte typing will be performed using an inflammatory Panel: e.g. CD4+ T cells, CD8+ T cells, CD19+ B cells, CD16+/CD56+ NK cells, CD4+/CD25+/CD127low regulatory T cells, CD45RA/CD45RO naive/memory T cells and activated immune cells.

OTHER OUTCOMES:
Adverse events | Baseline till 12 months after insertion of appliance
  Collection of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Corinna Lesley Seidel, Dr., Study Director — Department of Orthodontics and Orofacial Orthopedics; Lina Gölz, Prof.Dr., Study Director — Department of Orthodontics and Orofacial Orthopedics
Locations (1):
- Department of Orthodontics and Orofacial Orthopedics, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Seidel CL, Gerlach RG, Weider M, Wolfel T, Schwarz V, Strobel A, Schmetzer H, Bogdan C, Golz L. Influence of probiotics on the periodontium, the oral microbiota and the immune response during orthodontic treatment in adolescent and adult patients (ProMB Trial): study protocol for a prospective, double-blind, controlled, randomized clinical trial. BMC Oral Health. 2022 Apr 27;22(1):148. doi: 10.1186/s12903-022-02180-8. PMID 35477563